CLINICAL TRIAL: NCT05628909
Title: A Prospective, Randomized, Controlled, Multicentered Study of Vitrectomy With Silicone Oil Tamponade for Hypermyopic Foveoschisis.
Brief Title: Silicone Oil Tamponade for Vitrectomy of Hypermyopic Foveoschisis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Tongren Hospital (Other); Peking Union Medical College Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Henan Provincial People's Hospital (Other); Beijing Friendship Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Huaxi Hospital (Other); Shenzhen Eye Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Beijing Hospital (Other Government); Peking University Third Hospital (Other); Aier Eye Hospital, Beijing (Unknown); Peking University First Hospital (Other); Xuanwu Hospital, Beijing (Other); China-Japan Friendship Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Eye & ENT Hospital of Fudan University (Other); Zhongshan Ophthalmic Center, Sun Yat-sen University (Other); The Eye Hospital of Wenzhou Medical University (Other); Zhejiang Provincial People's Hospital (Other); The First People's Hospital of Xuzhou (Other); The First Affiliated Hospital of Dalian Medical University (Other); Second Hospital of Jilin University (Other); Xinjiang Production and Construction Corps Hospital (Unknown); The Affiliated Hospital of Inner Mongolia Medical University (Other); The Affiliated Hospital Of Guizhou Medical University (Other); Tianjin Medical University Eye Hospital (Other); Tianjin Medical University General Hospital (Other); Xinqiao Hospital of Chongqing (Other); Anhui Provincial Hospital (Other Government); Shengjing Hospital (Other); Lanzhou University Second Hospital (Other); The Fourth People's Hospital of Shenyang (Unknown); The Second Hospital of Hebei Medical University (Other); The Second Affiliated Hospital of Harbin Medical University (Other); The Affiliated Eye Hospital of Nanjing Medical University (Unknown); Second Xiangya Hospital of Central South University (Other); Shandong Eye Hospital (Other); Renmin Hospital of Wuhan University (Other); First Affiliated Hospital of Harbin Medical University (Other); Shanghai 10th People's Hospital (Other); Wuhan General Hospital of Guangzhou Military Command (Other); Southwest Hospital, China (Other); First Affiliated Hospital of Kunming Medical University (Other); First Hospital of China Medical University (Other); Wuxi People's Hospital (Other); The First Affiliated Hospital Of Southwest University, China (Unknown); Wuhan TongJi Hospital (Other); Shanghai Shi Bei Hospital (Unknown); Tianjin Eye Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Xi'an People's Hospital (Xi'an Fourth Hospital) (Other)
Responsible Party: Principal Investigator, Mingwei Zhao, Chief of Opthalmology department, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOME
Record Dates: First submitted 2022-11-08; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Hypermyopic Foveoschisis
MeSH Terms: interventions — Predictive Value of Tests

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Silicone oil group (Experimental): Patients randomized into this group were received pars plana vitrectomy surgery with silicone oil tamponade and without internal limiting membrane peeling. And silicone oil tamponade was removed at least 12 months after the primary surgery with completely resolved of foveoschisis.
  Interventions: Procedure: PPV with SO tamponade
- Gas group 1 (Active Comparator): Patients randomized into this group were received pars plana vitrectomy surgery with fovea-sparing internal limiting membrane peeling and gas tamponade.
  Interventions: Procedure: PPV with fovea-sparing ILMP and gas tamponade
- Gas group 2 (Active Comparator): Patients randomized into this group were received pars plana vitrectomy surgery with gas tamponade and without internal limiting membrane peeling.
  Interventions: Procedure: PPV with gas tamponade

INTERVENTIONS:
Procedure: PPV with SO tamponade — Patients randomized into silicone oil group were received pars plana vitrectomy surgery with silicone oil tamponade and without internal limiting membrane peeling. And silicone oil tamponade was removed at least 12 months after the primary surgery with completely resolved of foveoschisis.
  Arms: Silicone oil group
Procedure: PPV with fovea-sparing ILMP and gas tamponade — Patients randomized into gas group 1 were received pars plana vitrectomy surgery with fovea-sparing internal limiting membrane peeling and gas tamponade.
  Arms: Gas group 1
Procedure: PPV with gas tamponade — Patients randomized into gas group 2 were received pars plana vitrectomy surgery without internal limiting membrane peeling and gas tamponade.
  Arms: Gas group 2

SUMMARY:
The purpose of this study is to explore the efficiency and safety of the surgical procedure of pars plana vitrectomy with silicone oil tamponade and without internal limiting membrane peeling for myopic foveoschisis eyes with high risk of macular hole formation.

ELIGIBILITY:
Inclusion Criteria:

* patients with spherical ≥ -8 diopters or axial length ≥ 26.5mm.
* The foveoshisis combined with foveal detachment was showed on the OCT image. The foveal detachment height≥ 250 um ,and the thickness of sensory retina of foveal detachment was ≤100 um;
* patients signed the ICF.
* patients with BCVA ≤0.5,and with visual disturbance symptoms.

Exclusion Criteria:

* patients with macular hole
* accompanied or secondary of other fundus disease
* received vitrectomy due to other diseases
* glaucoma cannot be controled by medication
* patients with other retinal or choroidal disease that may affect VA
* poor patients compliance
* poor condition that cannot undertake the surgery
* optical opacities which make it difficult to exam fundus or measure on OCT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2022-10-29 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete resolved rate of foveoschisis observed on OCT image. | 18 months
  The compete resolved of foveoschisis was evaluated using OCT image.

SECONDARY OUTCOMES:
Best corrected visual acuity (BCVA) change compared with baseline BCVA. | 18 months
  Best corrected visual acuity (BCVA) change compared with baseline BCVA by ETDRS chart.
The posoperative macular hole formation rate. | 18 months
  The posoperative macular hole formation rate of different groups

CONTACTS AND LOCATIONS:
Overall Officials: Mingwei Zhao, M.D., Principal Investigator — Peking University People's Hospital; Yuou Yao, M.D., Study Director — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No